CLINICAL TRIAL: NCT04688281
Title: Spine Surgery for Adhesions in Patients Evaluated for Efficacy and Safety of MedicurtainⓇ Multicenter, Randomized, Evaluator-blind, Parallel-controlled Trial
Brief Title: Spine Surgery for Adhesions in Patients Evaluated for Efficacy and Safety of MedicurtainⓇ (Pivotal Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMT2011-SP-MC-03
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Intervertebral Disc Disorder; Thoracic Intervertebral Disc Disorders; Thoracolumbar Intervertebral Disc Disorders; Lumbosacral Intervertebral Disc Disorders; Tissue Adhesion, Surgery-Induced
Keywords: Medicurtain®; Sodium hyaluronate; Hydroxyethylstarch; Anti-adhesion barrier
MeSH Terms: conditions — Intervertebral disc disease; Tissue Adhesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUARDIX-SG® (Active Comparator): Treat GUARDIX-SG 5ml prefilled syringe after surgery
  Interventions: Device: GUARDIX-SG®
- Medicurtain® (Experimental): Treat Medicurtain® 5ml prefilled syringe after surgery
  Interventions: Device: Medicurtain®

INTERVENTIONS:
Device: Medicurtain® — Medicurtain® 5ml prefilled syringe
  Arms: Medicurtain®
Device: GUARDIX-SG® — GUARDIX-SG® 5ml prefilled syringe
  Arms: GUARDIX-SG®

SUMMARY:
This study was designed to evaluate the efficacy and safety of Medicurtain®, an antiadhesion barrier in patients who underwent In Situ Decompression for single level and unilateral herniated lumbar intervertebral disc. Subjects were randomly assigned either into Medicurtain® treatment group or control group. Adhesion formations between the two groups at 12 weeks after surgery were compared by using MRI-applied scar score, ODI (Oswestry Disability Index) and VAS.

DETAILED DESCRIPTION:
This study was multicenter, randomized, evaluator-blind, parallel-controlled trial. A subject aged between 20~70 years old who was reserved for In Situ Decompression for single level and unilateral herniated lumbar intervertebral disc considered to be eligible for study entry. Subject screening was conducted at Visit 1 (screening period) to determine study based on the results of the examination for the spine surgery. Subject who met the inclusion/exclusion criteria were randomly assigned into either the treatment and control group at Visit 2 (Baseline: 0day) and received the defined treatment according to the protocol.

Direct evaluation of the level of adhesion around surgical area was analyzed by measuring peridural fibrosis and scar score through MRI (Total MRI scar score). Jeffrey S. Ross et al. reported that in evaluating scar in disc region, MR has been used by many researchers and shows 96% accuracy in identifying scar in disc region. Also measuring the level of fibrosis in surgical wounds through MRI scar score has already been widely used in many large-scale studies and shows almost perfect conformity degree I inter-and intra-observer reading results.

Therefore based on literatures, this study measures the level of adhesion in surgical wounds through MRI scar score, which has been validated and widely used in similar studies. Using MRI 3 months after surgery, the level of scar in lumbar spinal column is evaluated. All MRI images should be evaluated by one radiologist unless the randomization of the treatment group and control group is revealed. Peridural fibrosis is evaluated on the improved and unimproved state of axial T1-weighted image contrast. In MR image evaluation, location of peridural fibrosis to 5 consecutive axial sections that are 4mm thick around the intervertebral disc is recorded; these 5 levels are divided into quadrant which are divided by 2 straight lines vertical to the center of thecal sac.

Degree of peridural fibrosis is scaled by scar grading scale in 0~4 point range according to the dimension of the quadrant filled with scar. Record the scar score of each quadrant of 5 levels (total of 20 grades-scar score method). The measured scar scores of the investigational device group and control device group are compared and evaluated with total of 20 scores on each quadrant of 5 levels (Total MRI score).

After 2 weeks (2 weeks±3days) of the index surgery, following tests were performed to evaluate the subject's condition and adverse events at before signing on the informed consent and after the surgery. The investigation device is composed of mainly Sodium Hyaluronate(HA) and Hydroxyethylstarch(HES) which were degraded in the liver and excreted from the kidney, therefore, it is included liver and kidney function test and blood coagulation test since abnormal function of blood coagulation can increase adhesion around the surgical wound area.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 ~ 70 years old
* Subject who is reserved with surgery for single-level or unilateral herniated lumbar Intervertebral disc
* Subject who is scheduled for In Situ Decompression(laparoscopic hysterectomy)
* Subject who does not respond to non-surgical treatment for at least past 6 weeks or require emergency surgery due to neural paralysis or excruciating pain
* Subject or his or her legal representative who signed and informed consent

Exclusion Criteria:

* Subject with multi-level or far lateral herniated lumbar intervertebral disc
* Subject with degenerative spinal disease or scoliosis
* Subject requires spinal fusion surgery
* Subject with severe liver or kidney disease
* Subject with lymph fluid or blood coagulation disease or medicated with blood clotting drug.
* Subject on oral or non-oral anti-diabetic drug or hypoglycemic drug
* Subject with suppressed immunity or autoimmune disease
* Subject with severe systemic disease
* Subject with infectious disease or healing disorder that may prevent normal healing process after surgery.
* Subject contraindicated with MRI scanning.
* Pregnant or lactating women
* Subject participated in other clinical trial within 30 days prior to the trial
* Subject justified not eligible to participate in the trial by Investigator

  * Subject undergone previous spinal surgery
  * Subject treated steroid epidural injection within 2 weeks or take oral steroid within 24 hours after surgery
  * Subject medicated aspirin or non-steroid anti-inflammatory drug within 7 days after surgery
  * Subject received myelogram or lumbar puncture within 24 hours after surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2013-03-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the average score of total MRI scar score evaluated by the independent evaluator after 12 weeks of the index surgery. | Week 12
  The intervertebral disc is divided into 5 consecutive axial sections and these 5 levels are divided into quadrant. Degree of peridural fibrosis is scaled by scar grading scale in 0~4 point range. (Total 20 score system)
  *Area of quadrant filled with scar: no scar = 0 point, 0%~25% = 1 point, 25%~50% = 2 point, 50%~75% = 3 point, 75%~100% = 4 point

SECONDARY OUTCOMES:
Comparison of the highest score of total MRI scar score evaluated by the independent evaluator after 12 weeks of the index surgery. | Week 12
  The intervertebral disc is divided into 5 consecutive axial sections and these 5 levels are divided into quadrant. Degree of peridural fibrosis is scaled by scar grading scale in 0~4 point range. (Total 20 score system)
  *Area of quadrant filled with scar: no scar = 0 point, 0%~25% = 1 point, 25%~50% = 2 point, 50%~75% = 3 point, 75%~100% = 4 point
Comparison of Oswestry Disability Index (ODI) final score for overall satisfaction with the surgery | Week 12
  The Oswestry Low Back Pain Disability Index (ODI) ODI Version 2.0 measure disability and quality of life in individuals with low back pain (LBP). It consists of questions related to Activities of Daily Living (ADLs) and pain, and is measured on a scale of 0-5 points for every 10 sections
Comparison of Visual Analog Scale (VAS) score for overall satisfaction with the surgery | Week 12
  The severity of pain was evaluated using a visual analogue scale (VAS). The participants were requested to put a line on the scale perpendicularly that matched to their pain intensity. VAS scores (0-100) represent the pain intensity as none, mild, moderate, or severe

OTHER OUTCOMES:
The incidence rate of adverse events | follow up to 12 weeks
  Safety and tolerability by collecting adverse events (AEs)
The incidence rate of treatment-emergent adverse event (TEAE) | follow up to 12 weeks
  Safety and tolerability by collecting treatment-emergent adverse event (TEAE)
The incidence rate of adverse device event | follow up to 12 weeks
  Safety and tolerability by collecting adverse device event (ADEs)
The incidence rate of serious adverse events | follow up to 12 weeks
  Safety and tolerability by collecting serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Suh Lee, MD, PhD, Principal Investigator — Samsung Medical Center, Gangnam-gu, Ilwon-dong 50, Seoul, South Korea; Eun-Sang Kim, MD, PhD, Principal Investigator — Samsung Medical Center, Gangnam-gu, Ilwon-dong 50, Seoul, South Korea; Ki-Tack Kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital, Gangdong-gu, Sangil-dong 149, Seoul, South Korea; Joomyung Kim, MD, PhD, Principal Investigator — Samsung Medical Center, Gangnam-gu, Ilwon-dong 50, Seoul, South Korea; Yong Cheol Yoon, MD, PhD, Principal Investigator — Hallym University Medical Center, Pyeongchon-dong 896, Anyang, Gyeonggi-do, South Korea; Bong-Soon Chang, MD, PhD, Principal Investigator — Seoul National University Hospital , Jongro-gu, Yeongeon-dong, Seoul, South Korea; Byung-Joon Shin, MD, PhD, Principal Investigator — Soonchunhyang University Hospital , Yongsan-gu, Daesagwan-ro 59, Seoul, South Korea
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, Ilwon-dong 50, South Korea

IPD SHARING:
Plan to Share IPD: No